CLINICAL TRIAL: NCT03894423
Title: Comprehensive CT Guided Coronary Bypass Graft Surgery
Brief Title: Comprehensive Computed Tomography Guidance of Coronary Bypass Graft Surgery
Status: Recruiting | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of California, San Diego (Other); VA Palo Alto Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Koen Nieman, Professor, Stanford University
Other Study IDs: IRB-49945; 1R01HL141712-01A1 (NIH); MZ-0048352 (Other: OnCore)
Record Dates: First submitted 2019-03-22; First posted 2019-03-28 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: CAD; Atheroscleroses, Coronary; Computed Tomography; Coronary Artery Bypass
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Apply CT angiography, CT perfusion imaging and advanced image processing techniques to improve revascularization decision-making and surgical strategies in patients undergoing coronary artery bypass graft surgery.

DETAILED DESCRIPTION:
The objective of this study is to integrate noninvasively acquired anatomical and functional information to develop clinically applicable tools for meaningful per-vessel revascularization decisions. The decisions will be based on quantitative lesion-specific ischemia and viability and flow simulations. These will be based on CT anatomy enhanced with a function for prediction of hemodynamic improvement after CABG.

Aim 1: Predict restoration of myocardial perfusion from coronary artery bypass graft surgery. The investigators will perform cardiac CT before and after CABG and measure absolute changes in myocardial perfusion as the functional outcome of CABG. The investigators will investigate clinical, surgical and imaging variables in association with post-CABG perfusion improvement on a per-vessel and per-patient level.

Aim 2: Non-invasively quantify vessel-specific ischemia for meaningful CABG decisions.

The investigators will develop and validate tools for assessment of vessel-specific ischemia and viability. The investigators will assess the potential impact of CT guided CABG by comparing the per-vessel need for grafting with standard care.

Aim 3: Predict CABG benefit through multi-parameter flow simulations Hypothesis: Integration of myocardial perfusion and viability can improve flow simulation models to predict CABG outcome. The investigators will develop new computational fluid dynamics models enriched with functional parameters and explore the potential of virtual grafting to improve hemodynamic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Planned elective CABG for coronary artery disease.
* CABG is the primary indication for surgery (but may include treatment of mild-moderate valvular disease).
* Age: ≥40 years.

Exclusion Criteria:

* Technical feasibility of the cardiac CT exams: redo-CABG, significant arrhythmia/mal-conduction, congenital conditions, severe valvular disease or cardiomyopathy (to the extent that the CT acquisition is technically challenged), inadequate understanding of the English language (to provide consent or follow instructions during the exams).
* Overall safety: unstable clinical condition (clinical heart failure, unstable angina, myocardial infarction <1 month prior).
* Radiation risk: pregnancy (cannot be ruled out), body weight >100kg.
* CT contrast medium-related: known allergy, renal failure
* Vasodilator related: known allergy, bronchial asthma requiring daily use of bronchodilators, Mobitz II or 3rd degree AV block, sick sinus node disease, clinically significant carotid artery narrowing, severe aortic stenosis or LVOT narrowing, systolic blood pressure below 90mmHg, (continued) use of dipyridamole or aminophylline.
* Inability to provide informed consent.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled to undergo coronary bypass graft surgery
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Change in myocardial blood flow from baseline measured by cardiac CT | 2 Months
  Myocardial blood flow will be measured by dynamic stress CT perfusion imaging before and 2 months after CABG. The primary endpoint is the difference MBF values between both examinations, per coronary distribution.

SECONDARY OUTCOMES:
Bypass graft obstruction by cardiac CT | 2 Months
  The presence of bypass grafts obstruction will be assessed on CT angiography
Change in angina pectoris assessed by SAQ | 1 Year
  Severity of anginal complaints will be assessed using the Seattle Angina Questionnaire before and 1 year after CABG.

CONTACTS AND LOCATIONS:
Overall Officials: Koen Nieman, MD, PhD, Principal Investigator — Stanford University
Locations (3):
- United States (3):
  - Palo Alto Veterans Affaird Healthcare System, Palo Alto, California
  - Stanford University, Palo Alto, California
  - University of California San Diego, San Diego, California

IPD SHARING:
Plan to Share IPD: No
No current plan to share data